CLINICAL TRIAL: NCT07175818
Title: Effects of Cold Plasma Systems Applied to PTFE and Silk Su-tures Used in Impacted Lower Third Molar Surgery on Post-operative Sequelae and Quality of Life
Brief Title: Cold Plasma-Treated Sutures in Third Molar Surgery: Effects on Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izzet Acikan (Other)
Responsible Party: Sponsor-Investigator, Izzet Acikan, Assistant Professor, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HRÜ/25.04.42
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Third Molars Extraction; Suture Materials
Keywords: third molar; Cold Plasma; PTFE; Silk

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- silk suture only (Active Comparator): The group in which only silk sutures will be used for wound closure after third molar extraction.
  Interventions: Procedure: Silk suture only
- PTFE suture only (Active Comparator): The group in which only PTFE sutures will be used for wound closure after third molar extraction.
  Interventions: Procedure: PTFE suture only
- silk suture and CAP (Experimental): The group in which cold atmospheric plasma is applied to silk sutures before wound closure with silk sutures after third molar extraction.
  Interventions: Procedure: Silk Suture + Cold athmospheric Plasma
- PTFE suture and CAP (Experimental): The group in which cold atmospheric plasma is applied to PTFE sutures before wound closure with PTFE sutures after third molar extraction.
  Interventions: Procedure: PTFE Suture + Cold athmospheric Plasma
- silk suture and CAP-Ar (Experimental): The group in which cold atmospheric argon plasma is applied to silk sutures before wound closure with silk sutures after third molar extraction.
  Interventions: Procedure: Silk Suture + Cold athmospheric argon Plasma
- PTFE suture and CAP-Ar (Experimental): The group in which cold atmospheric argon plasma is applied to PTFE sutures before wound closure with PTFE sutures after third molar extraction.
  Interventions: Procedure: PTFE Suture + Cold athmospheric argon Plasma

INTERVENTIONS:
Procedure: Silk suture only — After third molar extraction, the surgical wound will be closed using silk sutures without plasma application.
  Arms: silk suture only
Procedure: PTFE suture only — After third molar extraction, the surgical wound will be closed using PTFE sutures without plasma application.
  Arms: PTFE suture only
Procedure: Silk Suture + Cold athmospheric Plasma — After third molar extraction, silk sutures will be exposed to cold atmospheric plasma before being used for wound closure.
  Arms: silk suture and CAP
Procedure: PTFE Suture + Cold athmospheric Plasma — After third molar extraction, the surgical wound will be closed using PTFE sutures without plasma application.
  Arms: PTFE suture and CAP
Procedure: Silk Suture + Cold athmospheric argon Plasma — After third molar extraction, silk sutures will be exposed to cold atmospheric argon plasma before being used for wound closure.
  Arms: silk suture and CAP-Ar
Procedure: PTFE Suture + Cold athmospheric argon Plasma — After third molar extraction, PTFE sutures will be exposed to cold atmospheric argon plasma before being used for wound closure.
  Arms: PTFE suture and CAP-Ar

SUMMARY:
This study aims to compare the effectiveness of two types of surgical suture materials, silk and polytetrafluoroethylene (PTFE), used alone and in combination with cold atmospheric plasma systems, on postoperative outcomes such as pain, facial swelling, and limitation of mouth opening following mandibular third molar surgery. Written informed consent will be obtained from all volunteers prior to participation. For all groups, the surgical procedures will be performed on an outpatient basis under local anesthesia (2% lidocaine with 1:100,000 epinephrine) by a single surgeon. After achieving deep local anesthesia by blocking the inferior alveolar, buccal, and lingual nerves, the incision will be made using a modified envelope flap. Bone osteotomy will be performed under copious irrigation with sterile saline, using a high-speed straight surgical handpiece (20,000-40,000 rpm) and a #10 surgical round bur. After successful extraction of the teeth, bone margins will be appropriately smoothed, and the surgical site will be irrigated thoroughly with saline. The mucoperiosteal flap will then be closed with sutures according to the group criteria. For groups assigned to plasma application, plasma will be applied to the surface of the sutures. Pre- and postoperative evaluations will be conducted for all patients regarding facial swelling, limitation of mouth opening, and pain, using the same techniques. Assessment of swelling and mouth opening limitation will also be performed by the surgeon. Quality of life will be evaluated preoperatively and postoperatively for all participants. Follow-up examinations will be performed preoperatively, on the 2nd postoperative day, and on the 7th postoperative day. At these time points, facial scans will be recorded using the Qlone application on an iPhone 14, and STL files will be generated.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old and had no acute pericoronal infection

Exclusion Criteria:

* Individuals with systemic con-ditions such as diabetes mellitus, immunodeficiency, bleeding disorders, dyspepsia, or those classified as heavy smokers (over 10 cigarettes daily)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Assessment | Preoperative 20 minutes before local anesthesia administration, 1st. day, 2nd. day, 3rd. day, 4th. day, 5th. day, 6th. day, 7th. day.
  The patients' pain levels were evaluated using a 10-unit Visual Analog Scale (VAS). The patients were given a form on which they could mark the pain they felt as a score between 0 (no pain) and 10 (the most severe pain) at the following time points: 20 minutes before local anesthesia administration, and on postoperative day 1, day 2, day 3, day 4, day 5, day 6, and day 7. After completing these forms, the patients returned them at the end of the 7th day.
Facial Swelling Assessment | prior to surgery, on the second postoperative day, and on the seventh postoperative day
  Facial swelling was assessed by performing three-dimensional (3D) facial scans at three different time points: prior to surgery (T0), on the second postoperative day (T1), and on the seventh postoperative day (T2). All scans were obtained in the same clinical room under consistent lighting conditions. For image acquisition, the Qlone appli-cation (EyeCue Vision Technologies LTD.), compatible with iOS devices (iPhone 14, Apple Inc., CA, USA), was utilized, offering a guided face-scanning process. Upon completion, each scan was converted into an STL file, which was subsequently transferred to the 3D Slicer software. The paired scans were then superimposed, and volumetric differences were calculated.
Mouth Opening Assessment | prior to the operation, on the second postoperative day, and on the seventh postoperative day
  Interincisal mouth opening was measured both before and after surgery using a standard monoblock caliper. During the assessment, participants were seated upright with the orbitomeatal plane aligned parallel to the ground. The maximum unassisted midline in-terincisal distance was recorded in millimeters (mm) at three time points.
Quality of life Assessment | preoperatively, 2nd, and 7th days
  Quality of life was evaluated before and after surgery using the OHIP-14 questionnaire. Postoperative assessments were carried out on the preoperatively, 2nd, and 7th days following the procedure. Each question was rated on a 4-point scale: 1 = "never," 2 = "sometimes," 3 = "fairly often," and 4 = "very often." The possible total score ranged from 0 to 56, with higher scores reflecting greater impairment in quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam University, Faculty of Dentistry, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the results reported in the article, including anonymized demographic information, postoperative pain scores, swelling measurements, mouth opening values, and quality of life questionnaire results, will be shared. A data dictionary describing each variable will also be provided to ensure proper interpretation. Data will be made available upon reasonable request from qualified researchers after publication of the main results.
Supporting Information: ICF, Analytic Code

REFERENCES:
- [Background] Ercan UK, Ibis F, Dikyol C, Horzum N, Karaman O, Yildirim C, Cukur E, Demirci EA. Prevention of bacterial colonization on non-thermal atmospheric plasma treated surgical sutures for control and prevention of surgical site infections. PLoS One. 2018 Sep 5;13(9):e0202703. doi: 10.1371/journal.pone.0202703. eCollection 2018. PMID 30183745